CLINICAL TRIAL: NCT01432067
Title: Physical Activity Advices to Prevent Loss of Autonomy in Cancer Treated Elderly Patients. An Intervention Randomized Study
Acronym: CAPADOGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2010/23
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Cancer; Elderly Population
Keywords: cancer; geriatry; curative care; physical activity
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adaptated physical activity (Other): Physical activity advices adaptated to physical status of patients
  Interventions: Other: Adapted physical activity
- Standard physical activity (Other): Daily physical activities based on a standard guide
  Interventions: Other: Classic physical activities

INTERVENTIONS:
Other: Adapted physical activity — Physical activity advices according to a program adapted to physical status of the patient.
  Arms: Adaptated physical activity
Other: Classic physical activities — Daily physical activities based on a standard guide
  Arms: Standard physical activity

SUMMARY:
The investigators will propose to older cancer patients with good prognosis (curative care) a randomized trial of adapted physical activity during one year. To increase generalisation of the intervention the investigators intend to compare the PNNS advices (the French National Nutrition and Health Program) to a program targeted on the own capacities of each patient.

DETAILED DESCRIPTION:
Long-term evolution of successful-treated older patients is not well-known except for survival. They seem more affected by physical than psychological problems. The combined effects of aging, cancer, and treatments on muscle function could have hindered their usual physical activity. Cancer is associated with frailty. Fried and coll have defined a frailty phenotype as a combination of 3 or more of 5 conditions: exhaustion, loss of weight, decreased muscle strength, slow gait speed and low physical activity. Frail subjects have a higher risk of physical or cognitive disability and death. An intervention able to prevent frailty is of great interest for the older cancer patient and their quality of life. An intervention consisting of phone-program in physical activity has been associated with a decrease in self-reported disability in five-year obese survivors from cancer.

Patients will be randomized in two arms (1:1 ratio). Arm 1: Physical activity advices according to a program adapted to physical status of the patient assessed using SPPB (short physical performance battery) and the IPAQ questionnaire. A monthly phone support during one year will be performed by an adapted physical activity instructor and delivery of PNNS guide for subjects older than 55 y old. Arm 2: Delivery of PNNS guide for subjects older than 55 year old: recommendation of 1/2 hour physical activity of any kind.

Each patient will be followed during 2 years: First visit (V1) will take place before treatment. The subsequent visits will take place at 3 months (V2), 6 months (V3), 1 year (V4), 18 months (V5) and 2 years (V6), in which patients will complete questionnaires (IPAQ, QLQ-C30, one day dietary intakes), have clinical examinations (weight, performance status/ ECOG) and will be tested for physical facilities (SPPB, micro-fet2). These evaluations will be completed by the MMS / Fluency tests and the covered distance during 6 minutes at V1, V3, and V4.

ELIGIBILITY:
Inclusion Criteria:

* 70 years old or older
* Curative cares for cancer by chemotherapy and/ or surgery and/or hormonotherapy and/ or radiotherapy
* Patient with histologically proven lymphoma or carcinoma :

  * Colon, rectum or anal canal Cancer
  * Breast Cancer
  * Esophageal cancer
  * Otolaryngology Cancer
  * Kidney cancer
  * hepatocellular carcinoma
  * Stomach Cancer
  * Pancreatic cancer
  * Bile duct cancer
  * Ovarian Cancer
  * All lymphoma diffuse large B-cell and all peripheral T-cells lymphomas
  * All low-grade lymphoma: lymphocytes, lymphocytes and plasma cells, follicular, mantle, marginal zone (MALT and others)
  * Prostate cancer
  * Bladder Cancer
  * Lung cancer
  * adenocarcinoma of unknown primary origin compatible with previous quoted origin
* Performance status (ECOG) <4
* Patient who had given oral consent to participate in the study

Exclusion Criteria:

* Palliative cares for cancer

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 302 (Actual)
Dates: Start 2011-10-04 (Actual); Primary Completion 2016-06-10 (Actual); Study Completion 2016-06-10 (Actual)

PRIMARY OUTCOMES:
SPPB Score | 1 year
  The main outcome will be the proportion of subjects with a one-year decreased SPPB score of one point or more in 12.
Cognitive skills | 2 years
  MMS test, verbal fluency

SECONDARY OUTCOMES:
Quality of life | 2 years
  IPAQ, QLQ-C30, ADL, performance status (ECOG)
nutritional status | 2 years
Walking distance over 6 minutes | inclusion, 6 months and 1 year
isometric muscle strength measures of upper and lower limbs | 2 years
  microfet2 test
weight | 2 years
SPPB score | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle BOURDEL MARCHASSON, Pr, Principal Investigator — University Hospital, Bordeaux, France; Adélaïde DOUSSAU, Dr, Study Chair — University Hospital, Bordeaux, France
Locations (12):
- France (12):
  - CHU de Bordeaux - Hôpital Saint André, Bordeaux
  - Institut Bergonié, Bordeaux
  - CH de Dax, Dax
  - CHRU Lille, Lille
  - Centre Oscar Lambret, CLCC Lille, Lille
  - CHU de Limoges, Hôpital Dupuytren, Limoges
  - CH Mont de Marsan, Mont-de-Marsan
  - CHU Bordeaux - hôpital Xavier Arnozan, Pessac
  - Institut jean Godinot, CLCC Reims, Reims
  - Centre hospitalier de Senlis, Senlis
  - Centre Alexis Vautrin CLCC Nancy, Vandœuvre-lès-Nancy
  - CHU Nancy hôpital adulte du brabois, Vandœuvre-lès-Nancy